CLINICAL TRIAL: NCT03887143
Title: National Retrospective Study Of Recanalization Treatments In Pediatric Arterial Ischemic Stroke (Intra-venous Thrombolysis and/or Endovascular Treatment: Thrombectomy, Intra-arterial Thrombolysis)
Brief Title: National Retrospective Study Of Recanalization Treatments In Pediatric Arterial Ischemic Stroke
Acronym: KID-CLOT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI18025HLJ
Record Dates: First submitted 2019-01-10; First posted 2019-03-22 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Arterial Ischemic Stroke
Keywords: Ischemic stroke; children; recanalization treatment; thrombolysis; thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arterial ischemic stroke in patients less than 18 years old: Patients < 18 years old
  * Suspected or confirmed cerebral infarction
  * With recanalization treatment in the acute phase: intra-venous thrombolysis +/- intra-arterial thrombolysis +/- thrombectomy
  * Patients treated between January 2015, 1st and May 2018, 31st

SUMMARY:
The purpose of this study is to evaluate recanalization treatments use, safety and efficacy at the acute phase of arterial ischemic stroke in pediatric patients

DETAILED DESCRIPTION:
Arterial ischemic stroke outcomes benefited from the implementation of recanalization treatments (IV thrombolysis, endovascular treatments) and adapted management pathways in adult patients. Nevertheless randomized trials did not enroll patients under the age of 18 years old and data concerning these treatments in children are scarce. As it is much less frequent than in adults, recognition of stroke is often delayed in children. Consequently, acute phase trials are difficult to set up and perform. The phase I multicentric international prospective trial TIPS (Thrombolysis in Pediatric Stroke) was prematurely stopped because of poor enrollment. Published retrospective regional (Paris-Ile-de-France region, France) and national (Switzerland) studies addressed the feasibility of such treatments but, because of small samples (less than 20 patients in each study), efficiency and prognostic factors could not be addressed.

Exhaustive retrospective studies in a definite geographic area but with a sufficient number of patients in a limited inclusion period would provide these crucial data and address these questions with good relevance and limited bias.

ELIGIBILITY:
Inclusion Criteria:

* Patients under 18 years old
* Suspected or confirmed cerebral infarction
* With recanalization treatment in the acute phase : intravenous thrombolysis +/- intra-arterial thrombolysis +/- thrombectomy
* Patients treated between the January 2015, 1st and the May 2018, 31st
* Collection of non-opposition from legal representatives

Exclusion Criteria:

- Refusal of the patient's legal representative to participate in the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged less than 18 yo with arterial ischemic stroke and recanalization treatment at the acute phase, treated in France during the study period. Sample recruited from pediatric and adult databases of child neurology, stroke, and interventional radiology units
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Acute management of stroke: | 1 day
  Median time from symptom onset to Imaging (minutes)
Acute management of stroke: | 1 day
  Median time from symptom onset to beginning of recanalization treatment (minutes)
Acute management of stroke: | 1 day
  Median door-to-needle delay (minutes)

SECONDARY OUTCOMES:
Treatment-emergent adverse events: | 7 days
  Intracranial hemorrhage (yes/no)
Treatment-emergent adverse events: | 7 days
  clinically symptomatic (yes/no)
Treatment-emergent adverse events: | 7 days
  Peripheral hemorrhage (yes/no)
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  age of onset (year, months)
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  Mechanism of stroke (CASCADE classification)
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  stroke location (name of artery territory)
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  time from symptom onset to beginning of recanalization treatment (minutes)
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  initial imagine ASPECT Alberta Stroke Program Early CT Score. score (units on an scale). The ASPECTS score is a 10-point quantitative topographic CT scan score used in patients with middle cerebral artery (MCA) stroke. I has also been adapted to be used with MR scans.
  All scale ranges : Segmental assessment of the MCA vascular territory is made and 1 point is deducted from the initial score of 10 for every region involved (caudate, putamen, internal capsule, nsular cortex, M1(anterior MCA cortex=frontal operculum), M2(MCA cortex lateral to insular ribbon=anterior temporal lobe), M3(posterior MCA cortex=posterior temporal lobe, M4(anterior MCA territory immediately superior to M1), M5(lateral MCA territory immediately superior to M2), M6(posterior MCA territory immediately superior to M3)
  For each scale, values better or worse :
  In adults, an ASPECTS score less than or equal to 7 predicts a worse functional outcome at 3 months as well as symptomatic hemorrhage
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  Association with :Modified Rankin Scale - mRS (Units on a scale)The mRS is a 6-point quantitative measure of functional independence.
  All scale ranges:
  0=No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance disability; requiring some help, but able to walk without assistance
  3. Moderate
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
  For each scales range, values better or worse :
  In the literature, good outcome is usually considered for patients with mRS [0-2]. Very good outcome is considered for patients with mRS [0-1]. We will use the same thresholds
factors potentially associated with clinical outcome: univariate and multivariate analysis, step by step analysis | 12 months
  Association with :
  - The Pediatric Stroke Outcome Measure - PSOM (Units on a scale) =scale has been designed and published to quantify functional consequences of stroke in children. The PSOM is a detailed neurological examination, with outcome scored in terms of degree of impairment in each of language, cognition, and sensorimotor. We wil use the PSOM-SNE version (PSOM-Short Neuro Exam version).
  All scale ranges (0-0,5-1 or 2):
  - Sensorimotor deficit, Language Deficit - Production, Language Deficit - Comprehension, Cognitive or Behavioural Deficit. Total score on 10
  For each scale range, values better or worse:
  Total impairment scores (out of a maximum of 10) will be considered as previously published, i.e. total score 0 or 0.5 representing good outcome, and poor outcome ≥1.
  All subscales ranges (Normal, Anormal, Not Done):
  Level of consciousness, Behaviour, mental status, Language, Cranial nerves, Motor testing, Tendon reflexes, Fine motor coordination, Sensory, Gate

CONTACTS AND LOCATIONS:
Overall Officials: Manoelle Kossorotoff, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker- Enfants Malades Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kossorotoff M, Kerleroux B, Boulouis G, Husson B, Tran Dong K, Eugene F, Damaj L, Ozanne A, Bellesme C, Rolland A, Bourcier R, Triquenot-Bagan A, Marnat G, Neau JP, Joriot S, Perez A, Guillen M, Perivier M, Audic F, Hak JF, Denier C, Naggara O; KidClot Group. Recanalization Treatments for Pediatric Acute Ischemic Stroke in France. JAMA Netw Open. 2022 Sep 1;5(9):e2231343. doi: 10.1001/jamanetworkopen.2022.31343. PMID 36107427
- [Derived] Tudorache R, Kossorotoff M, Kerleroux B, Denier C, Naggara O, Boulouis G; KID-CLOT Group. Determinants of Timely Access to Recanalization Treatments and Outcomes in Pediatric Ischemic Stroke. Stroke. 2024 Nov;55(11):2716-2719. doi: 10.1161/STROKEAHA.124.046417. Epub 2024 Oct 1. PMID 39351662
- See also: Related Info — http://www.chu-st-etienne.fr/avcpediatrie